CLINICAL TRIAL: NCT05375084
Title: A Phase 1 Study of the SHP2 Inhibitor BBP-398 (Formerly Known as IACS-15509) in Combination With the Programmed Death Receptor-1 Blocking Antibody Nivolumab in Patients With Advanced Non-Small Cell Lung Cancer With a KRAS Mutation
Brief Title: SHP2 Inhibitor BBP-398 in Combination With Nivolumab in Patients With Advanced Non-Small Cell Lung Cancer With a KRAS Mutation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Navire Pharma Inc., a BridgeBio company (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NAV-1004
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Non Small Cell Lung Cancer; Solid Tumor
Keywords: KRAS mutation; MAPK-pathway alterations; NSCLC; SHP2
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation Level 1 (Experimental): Level 1 oral capsules administered in combination with nivolumab
  Interventions: Drug: BBP-398 with nivolumab
- Dose Escalation Level 2 (Experimental): Level 2 oral capsules administered in combination with nivolumab
  Interventions: Drug: BBP-398 with nivolumab
- Dose Escalation Level 3 (Experimental): Level 3 oral capsules administered in combination with nivolumab
  Interventions: Drug: BBP-398 with nivolumab
- Dose Expansion (Experimental): RP2D defined dose. Oral capsules administered in combination with nivolumab
  Interventions: Drug: BBP-398 with nivolumab

INTERVENTIONS:
Drug: BBP-398 with nivolumab — BBP-398 administered orally once a day (QD); nivolumab administered intravenously every 4 weeks (Q4wks)

SUMMARY:
This is a Phase 1 study of BBP-398, a SHP2 inhibitor, in combination with nivolumab, a PD-1 antibody, in patients with NSCLC with a KRAS mutation. The study involves 2 parts: Phase 1a Dose Escalation and Phase 1b Dose Expansion.

DETAILED DESCRIPTION:
The primary objective for Phase 1a Dose Escalation is to evaluate the safety, tolerability, and RP2D of BBP-398, a SHP2 inhibitor, when used in combination with nivolumab in patients with advanced NSCLC with a KRAS mutation who have failed standard of care treatment.

The primary objective for Phase 1b Dose Expansion is to evaluate the antitumor activity of BBP-398, as defined by the ORR (per investigator) according to RECIST v1.1, when used in combination with nivolumab in patients with advanced NSCLC with a KRAS mutation who have failed standard of care treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients must have histologically documented, locally advanced and unresectable, or metastatic NSCLC with documentation of a KRAS mutation within the 1 year prior to screening.
* Patients must have measurable disease by RECIST v1.1.
* Patients must have a minimum life expectancy of >12 weeks after start of study treatment.
* Patients must have progression or disease recurrence on or after at least one prior line of systemic therapy, which must include platinum-based doublet chemotherapy and anti-PD-(L)1 therapy.
* Patients must have experienced progressive or recurrent disease occurring either during treatment or within 90 days after discontinuing anti-PD-(L)1 therapy.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
* Patients must have adequate organ function.

Key Exclusion Criteria:

* Patients that have participated in an interventional clinical study within the last 4 weeks.
* Patients that have received radiotherapy or proton therapy with a limited field of radiation for palliation within 1 week of the start of study treatment, OR radiation to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the start of study treatment.
* Patients with known central nervous system (CNS) tumors or active CNS metastases.
* Patients that have experienced progressive disease (PD) within the first 120 days of initiating treatment with an anti- PD-(L)1 agent (e.g., primary refractory).
* Patients that have a history of allogenic bone marrow transplant.
* Patients that have select known or suspected autoimmune disease.
* Patients that have a condition requiring systemic treatment with either corticosteroids (>10 mg prednisone equivalent) or other immunosuppressive medication within 14 days of study start.
* Patients that have received any live/attenuated vaccine within 30 days of first study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Phase 1a Dose Escalation: Assess safety, tolerability, and recommended phase 2 dose (RP2D) of BBP-398 in combination with nivolumab | Completion of 1 Cycle (28 days)
Phase 1b Dose Expansion: Assess antitumor activity of BBP-398 in combination with nivolumab | Completion of 1 Cycle (28 days)
  Anti-tumor activity will be defined by objective response rate (ORR) according to RECIST v1.1

SECONDARY OUTCOMES:
Assess preliminary antitumor activity of BBP-398 in combination with nivolumab | Completion of 1 Cycle (28 days)
  Anti-tumor activity will be defined by objective response rate (ORR) [escalation], duration of response (DOR) and progression free survival (PFS), as defined by RECIST v1.1. and overall survival (OS) [both escalation and expansion]
Phase 1b Dose Expansion: Assess safety and tolerability of BBP-398 at the RP2D, in combination with nivolumab | Completion of 1 Cycle (28 days)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Highlands Oncology, Springdale, Arkansas
  - Scripps Clinic Torrey Pines, La Jolla, California
  - Providence Medical Foundation, Santa Rosa, California
  - Memorial Regional Hospital (Memorial Cancer Institute), Hollywood, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - University of Pennsylvania (Abramson Cancer Center), Philadelphia, Pennsylvania
  - Medical University of South Carolina (MUSC) - Hollings Cancer Center, Charleston, South Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - Millennium Research and Clinical Development, Houston, Texas
  - NEXT Oncology, Fairfax, Virginia